CLINICAL TRIAL: NCT00426426
Title: A Randomised Controlled Trial Comparing the Effectiveness of Cognitive Behaviour Therapy (CBT) With Metacognitive Therapy (MCT) in the Treatment of Patients With Generalised Anxiety Disorder (GAD)
Brief Title: Comparing Cognitive Behaviour Therapy (CBT) With Metacognitive Therapy (MCT) in the Treatment of GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Penn State University (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 4.2006.2369; NSD: sak 15436 (Other: NSD)
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meta-Cognitive Therapy (Active Comparator): first Meta-cognitive therapy then Cognitive Behaviour Therapy
  Interventions: Behavioral: Cognitive-Behavioural Therapy; Behavioral: Meta-Cognitive Therapy; Behavioral: Waiting list
- Cognitive Behaviour Therapy (Active Comparator): first Cognitive Behaviour Therapy then Meta-cognitive therapy
  Interventions: Behavioral: Cognitive-Behavioural Therapy; Behavioral: Meta-Cognitive Therapy; Behavioral: Waiting list
- Waiting List (Other): Waiting List
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: Cognitive-Behavioural Therapy — 12 sessions with Cognitive-Behavioural Therapy (CBT), and waiting list will be over 12 weeks, and then allocated into Meta-Cognitive Therapy.
  Arms: Cognitive Behaviour Therapy; Meta-Cognitive Therapy
Behavioral: Meta-Cognitive Therapy — 12 sessions with Meta-Cognitive Therapy (MCT), and waiting list will be over 12 weeks, and then allocated into Cognitive-Behavioural Therapy .
  Arms: Cognitive Behaviour Therapy; Meta-Cognitive Therapy
Behavioral: Waiting list

SUMMARY:
Meta Cognitive Therapy (MCT) has been introduced as a new specific treatment for generalised anxiety disorder. So far, no studies have examined CBT and MCT in comparison with each other in a randomised controlled trial. Sixty patients with a diagnosis of generalised anxiety disorder will be selected and randomised into three treatment conditions. The first group (N=20) will be treated with CBT, the second group (N=20) with MCT, and the third condition is a waiting list control (N=20). The patients in both groups will have full treatment, in accordance to treatment manuals developed by the originators. Patients in the waiting list control will be randomly allocated to either CBT or MCT after 12 weeks of waiting period.

The patients will be assessed with the primary measures at pre-treatment, at the end of treatment, and at follow-up after one and two years. In addition they will be assessed weekly on symptom measures and worry outcome diary. The therapist will be treating equally amount of patients in both conditions to control for any biased distribution connected to the therapist's characteristics.

Measures will be used on at least three main sources; self-report inventories (including symptom diaries), clinical assessments by independent raters and psycho-physiological assessments.

We aim to (1) evaluate and compare the effectiveness of CBT and MCT, (2) investigate the patterns of change and the mechanisms of action involved during treatment in each of the conditions and, (3) evaluate pre and post-treatment somatic change by psycho-physiological assessments as a response to CBT and MCT.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to entry in the study.
2. Diagnosed with generalised anxiety disorder (DSM-IV, APA, 1994).
3. 18 years or older.

Exclusion Criteria:

1. Known somatic diseases
2. Psychosis
3. Past suicidal attempts and/or current intent
4. PTSD
5. Cluster A or cluster B personality disorder
6. Substance dependence
7. Not willing to accept random allocation.
8. Patients not willing to withdraw psychotropic medication for a period of 4 weeks prior to entry to the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PSWQ by post treatment and by two year follow up. | March 2011
STAI-T | March 2011

CONTACTS AND LOCATIONS:
Overall Officials: Leif E Kennair, PhD, Principal Investigator — Dept. of Psychology, NTNU; Hans M Nordahl, Ph.D, Study Director — Department of Psychology
Locations (1):
- Department of Psychology, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Johnson SU, Hoffart A, Nordahl HM, Wampold BE. Metacognitive therapy versus disorder-specific CBT for comorbid anxiety disorders: A randomized controlled trial. J Anxiety Disord. 2017 Aug;50:103-112. doi: 10.1016/j.janxdis.2017.06.004. Epub 2017 Jun 15. PMID 28651207
- [Result] Nordahl HM, Borkovec TD, Hagen R, Kennair LEO, Hjemdal O, Solem S, Hansen B, Haseth S, Wells A. Metacognitive therapy versus cognitive-behavioural therapy in adults with generalised anxiety disorder. BJPsych Open. 2018 Sep 11;4(5):393-400. doi: 10.1192/bjo.2018.54. eCollection 2018 Sep. PMID 30294448